CLINICAL TRIAL: NCT01714297
Title: A Prospective Randomized, Double Blind Study to Evaluate Safety and Effect With Pre Versus Postoperative Start of Thromboprophylaxis With Dalteparin
Brief Title: Preoperative Versus Postoperative Start With Thromboprophylaxis in THA (Total Hip Arthroplasty)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Pål Borgen, MD, MD., Vestre Viken Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REK Sør-øst s-08012d
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Arthritis of the Hip; Transfusion Related Complications; Infection; Wound Discharge
Keywords: cemented total hip arthroplasty; blood loss; wound discharge; thromboprophylaxis; biomarkers
MeSH Terms: conditions — Infections; Hemorrhage | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dalteparin 5000IU s.c. (Active Comparator): 5000IU dalteparin s.c. injected the evening before cemented total hip arthroplasty
  Interventions: Drug: dalteparin 5000 IU s.c.
- saline (Placebo Comparator): Syringes of Saline with the same volume as in the dalteparin injections are injected the evenings before total hip arthroplasty. Dalteparin 5000IU are injected 6 hours after surgery and the concomitant 33 days
  Interventions: Drug: dalteparin 5000 IU s.c.

INTERVENTIONS:
Drug: dalteparin 5000 IU s.c. — All patients receive injections with either 5000IU dalteparin or saline in the same volume the evening before surgery. All patients receive 5000IU dalteparin 6 hours after surgery and every day from day 2 until day 35.
  Other Names: Fragmin

SUMMARY:
The purpose of this study is to determine if there are differences in clinical events, i.e bleeding with associated morbidity, if thromboprophylaxis with LMWH (Low Molecular Weight Heparin) is initiated before or after surgery.

ELIGIBILITY:
Inclusion Criteria:

-patients 50 years or older undergoing cemented total hip arthroplasty for primary osteoarthritis

Exclusion Criteria:

* allergy to Low-Molecular-Weight -Heparin
* bleeding disorders
* renal failure
* hepatic disease
* active treatment for malignancy
* history of deep venous thrombosis or pulmonary embolism
* major operations,trauma,stroke or cardiac infarction the last 3 months before surgery.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
total blood loss | during and after surgery
  measured blood loss during surgery and in wound drains

SECONDARY OUTCOMES:
transfusion requirements | during and after surgery
  number of units packed red blood cells
incidence of bleeding events | during and after surgery
  excessive bleeding, wound hematoma, wound secretion, other bleeding events
other complications | during and after surgery
  all other complications related to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olav Reikeras, MD, Phd, Study Chair — Oslo University Hospital
Locations (1):
- Martina Hansen's Hospital, Sandvika, Gjettum, Norway

REFERENCES:
- [Result] Borgen PO, Dahl OE, Reikeras O. Blood loss in cemented THA is not reduced with postoperative versus preoperative start of thromboprophylaxis. Clin Orthop Relat Res. 2012 Sep;470(9):2591-8. doi: 10.1007/s11999-012-2320-9. Epub 2012 Apr 3. PMID 22476844